CLINICAL TRIAL: NCT02907528
Title: Furcation Therapy With Enamel Matrix Derivative: Effects on the Subgingival Microbiome
Brief Title: Furcation Therapy With Enamel Matrix Derivative
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Purnima Kumar, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OSU-FAPESP 101
Record Dates: First submitted 2016-09-11; First posted 2016-09-20 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BONE Group (Placebo Comparator): bone substitute consisting of beta tricalcium phosphate/hydroxyapatite (βTCP/HA- Bone Ceramic® Straumann, Basel, Switzerland)
  Interventions: Biological: Bone
- BONE+EMD Group (Active Comparator): mixture of enamel matrix derivative proteins (EMD) (Emdogain® Straumann, Basel, Switzerland) and bone substitute consisting of βTCP/HA (Bone Ceramic® Straumann, Basel, Switzerland);
  Interventions: Biological: Bone; Biological: EMD
- EMD Group (Experimental): enamel matrix derivative (EMD - Emdogain® Straumann, Basel, Switzerland)
  Interventions: Biological: EMD

INTERVENTIONS:
Biological: Bone — Furcation defect regenerated with bone graft material
  Arms: BONE Group; BONE+EMD Group
Biological: EMD — Furcation defect regenerated with EMD
  Arms: BONE+EMD Group; EMD Group

SUMMARY:
Objective: To clinically evaluate mandibular furcation treated with Beta tricalcium phosphate/hydroxyapatite (βTCP/HA) isolated or combined with enamel matrix derivative (EMD + βTCP/HA) and EMD alone.

Material and Methods: 39 patients, presenting at least one mandibular class II furcation defect, probing pocket depth (PPD) ≥ 4 mm and bleeding on probing, were included. The defects were assigned to the βTCP/HA group 1 (n = 13); open-flap debridement (OFD) + βTCP/HA filling; βTCP/HA + EMD group 2 (n = 13); OFD + βTCP/HA + EMD filling; and EMD group 3 (n = 13) OFD + EMD filling. Plaque (PI) and gingival index (GI), PPD, relative gingival margin position (RGMP), vertical and horizontal attachment level (RVCAL and RHCAL), and furcation diagnosis were evaluated at baseline, 6 and 12 months.

DETAILED DESCRIPTION:
Although enamel matrix derivative (EMD) has been used to promote periodontal regeneration, little is known of its effect on the microbiome. Therefore, this investigation aimed to identify the changes in periodontal microbiome following treatment with EMD using a deep-sequencing approach. Thirty-nine patients having mandibular class II buccal furcation defects were randomized to beta-tricalcium-phosphate/hydroxyapatite graft (BONE group), EMD+BONE or EMD alone. Plaque was collected from furcation defects at baseline, 3 and 6 months post-treatment. Bacterial DNA was analyzed using terminal restriction fragment length polymorphism (t-RFLP) and 16S pyrotag sequencing. 169,000 classifiable sequences were compared to HOMD using the QIIME and PhyloToAST pipelines. Statistical comparisons were made using parametric tests. At baseline, a total of 422 species were identified from the 39 defects, belonging to Fusobacterium, Pseudomonas, Streptococcus, Filifactor and Parvimonas. All three regenerative procedures predictably altered the disease-associated microbiome, with a restitution of health-compatible species. However, EMD and BONE+EMD groups demonstrated more long-term reductions in higher number of species than in BONE group (p<0.05), especially disease-associated species e.g. Selenomonas noxia, F.alocis, and Fusobacterium. EMD may promote periodontal regeneration by predictably altering a dysbiotic subgingival microbiome, decreasing pathogen richness and increasing commensal abundance.

ELIGIBILITY:
Inclusion Criteria:

* Untreated ChronicPeriodontitis

Exclusion Criteria:

* Diabetes Pregnancy Current Smoking

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Shifts in the subgingival microbiome at 3 and 6 months in response to the interventions | 6 months
  Subgingival microbial plaque samples will be collected at baseline and at the 3 and 6-month re-evaluation visits. Bacterial samples will be removed from the paper points by adding 200µl of phosphate buffered saline (PBS) and vortexing for 1 minute. The paper points were then removed, and DNA isolated using a Qiagen MiniAmp kit (Valencia, CA) according to the manufacturer's instructions. Multiplexed bacterial tag-encoded FLX amplicon pyrosequencing will be performed using the Titanium platform. High quality, classifiable sequences (quality score >25, >200bp length) were clustered into species-level operational taxonomic units (s-OTUs) at 97% sequence similarity and assigned a taxonomic identity by alignment to the HOMD database using the Blastn algorithm. Primary outcome measures will be changes in diversity, equitability and levels of pathogens.

CONTACTS AND LOCATIONS:
Overall Officials: purnima Kumar, Principal Investigator — Ohio State University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Queiroz LA, Casarin RCV, Dabdoub SM, Tatakis DN, Sallum EA, Kumar PS. Furcation Therapy With Enamel Matrix Derivative: Effects on the Subgingival Microbiome. J Periodontol. 2017 Jul;88(7):617-625. doi: 10.1902/jop.2017.160542. Epub 2017 Mar 17. PMID 28304211